CLINICAL TRIAL: NCT06703762
Title: Efficacy of Photobiomodulation on Wound Healing and Il-6 in Neuropathic Foot Ulcer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatma Mahmoud Abd Allah Abd Alsadek, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005252
Record Dates: First submitted 2024-11-20; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Neuropathic Foot Ulcer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- He-Ne low level laser (LLL) + Conventional traditional treatment (Experimental): It will include 34 patients with chronic neuropathic foot ulcer from both sex. They will receive He-Ne LLL for chronic neuropathic foot ulcer with pulsed wave form, visible ray, wave length of 632.8 nm, peak potency of 30 mW, (Laser -HTM). The application time will be 80 (4 J/cm2) seconds. The application will be 3 sessions /week for 4 weeks on the sole of the foot + Conventional traditional treatment.
  Interventions: Other: He-Ne low level laser (LLL); Other: Conventional traditional treatment
- Conventional traditional treatment (Active Comparator): It will include 34 patients with chronic neuropathic foot ulcer from both sex. They will receive conventional traditional treatment (regular sharp debridement of calluses surrounding the ulcer, use of walking or total-contact casts for off-loading and regular moist dressing patients will be instructed to use only sodium chloride (saline solution 0.9%), regarding the daily asepsis of the ulcer).
  Interventions: Other: Conventional traditional treatment

INTERVENTIONS:
Other: He-Ne low level laser (LLL) — Patients in the experimental group will receive treatment with LLLT. The ulcer bed will be irradiated locally with red light (660 nm). The ulcer size and its depth will be used as the basis to calculate the duration of exposure needed to deliver 3-10 J/cm² for 15 to 20 minutes. The application will take place in 3 sessions per week for 4 weeks. Each patient will be asked to lie in a supine position with the ulcer easily exposed to the laser beam, and they will be instructed to wear laser glasses and avoid looking directly at the beam until the end of the session.
  Arms: He-Ne low level laser (LLL) + Conventional traditional treatment
Other: Conventional traditional treatment — All patients in both the groups will receive the required, conventional treatments of diabetic wound care, including dressing, antibiotics, controlling diabetes, cholesterol, and blood pressure along with aggressive drug treatment and wound debridement when needed.

SUMMARY:
The aim of this study is to detect the effect of Laser Photobiomodualation on the wound healing and Il-6 in neuropathic foot ulcer.

DETAILED DESCRIPTION:
Wound healing is a complex, interactive, and integrative event, involving cellular and chemotactic activity with release of chemical mediators associated with vascular responses and cell proliferation. It consists in a sequence of events leading to the closure of dermal injuries. The repair follows steps of inflammation, re-epithelization, wound contraction, and matrix remodeling. The healing process can be influenced by various local and systemic factors.

The ulcer treatment in the diabetic foot requires a multidisciplinary approach, including revascularization and surgical procedures, as well as the infection treatment, physiotherapeutic rehabilitation with electric phototherapeutic resources to control edema, pain, metabolic disorders, tissue malnutrition, co morbidities, precise treatment of the wound and biomechanics' decompression that will help in amputation prevention.

Biophotomodulation in the form of Low level laser (LLL) irradiation can promote cell migration and cell proliferation by stimulating mitochondrial activity and maintaining viability without causing damage to the wounded cells.

The usage of LLLT presents itself as being a new therapeutic proposal, seeking the cure of these injuries, the improvement on the quality of life of the affected individuals, as well as the reduction of the costs of the treatment in the health system, this study aims to identify the effects of low-level laser therapy on neuropathic foot ulcer healing and the effect of LLL on the hyperglycemic-induced inflammatory response in IL-6 and sought to identify which pathway it might achieve this effect.

ELIGIBILITY:
Inclusion Criteria:

* All patient will be diagnosed with neuropathic foot ulcer.
* All patient diagnosed as type II Diabetes Mellitus.
* Wound size a 6-12 cm2.
* Diabetic ulcers will be in grade 2 and 3 (Partial thickness skin loss involving epidermis and or dermis (superficial, abrasion, blister, and / or full thickness skin loss damage ore necrosis of subcutaneous tissue may extend down to but not through underlying fascia.

Exclusion Criteria:

* Presence of osteomyelitis.
* Patients associated with critical illness who needs intensive care.
* Patients who suffer from cellulitis.
* Patients who suffer from nerve injury.
* Pregnancy.
* Smokers
* Malignant diseases
* Use of immunosuppressive drugs
* Phenytoin, cyclosporine, calcium channel blockers, etc.
* Patients who not have burn or ulcer or trauma in this area

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-11-26 (Estimated); Primary Completion 2025-01-26 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of Ulcer Length | 4 weeks
  The length of the ulcer can be precisely measured using the Imito Measure application. By utilizing a specialized marker for calibration, the app allows users to trace the ulcer's longest dimension. After capturing an image, the app calculates the length automatically, providing an accurate measurement.
Measurement of Ulcer Width | 4 weeks
  The width of the ulcer is measured in a similar manner using the Imito Measure app. Users trace the widest part of the wound, and the app, after calibration with the marker, determines the exact width from the captured photo.
Measurement of Ulcer Area | 4 weeks
  The area of the ulcer is calculated by encircling the entire wound boundary using the Imito Measure application. The app uses the calibration marker to ensure accuracy and then automatically computes the total wound area. The Imito Measure application has been scientifically validated as a reliable alternative to traditional wound measurement methods, such as wound rulers.
Measurement of volume of the ulcer | 4 weeks
  It can be measured by using Syringe method by injecting saline into the wound until it overflows from the wound and measure the amount of saline.
Assessment of serum IL-6 level | 4 weeks
  Samples of venous blood from the cubital vein will be taken from each patient. Collected blood samples will be transferred into a test tube pre-fabricated with an anticoagulant. The blood samples will remain in the test tubes for about 30 minutes and will then be distributed to a biochemical laboratory, where they will be centrifuged at 6,000 rpm for 10 minutes. The serum will be separated from the test tube and transferred to an Eppendorf tube. All serum samples will be stored at -80°C until complete analysis and measurement of IL-6 levels. The IL-6 level in the serum will then be determined. Additionally, fasting blood sugar levels will be measured to assess the stabilization of the condition.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Mohamed Abd El-baky, PhD, Study Chair — Professor, Cairo university
Locations (1):
- Cairo University, Giza, Egypt